CLINICAL TRIAL: NCT05783284
Title: HS2 US Liver Reader Study
Status: Completed | Type: Observational
Sponsor: HoloCare AS (Industry)
Responsible Party: Sponsor
Other Study IDs: CIHS2-002
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Reader Study
Keywords: Holographic visualization

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Readers: 5 trained GI surgeons within liver surgery (the readers) will identify pre-defined anatomical landmarks in liver CT images that have been processed by HS2
  Interventions: Device: Holocare Studio 2 (HS2)

INTERVENTIONS:
Device: Holocare Studio 2 (HS2) — 3D HV

SUMMARY:
The purpose of this study is to to assess the ability of 5 Gastro-Intestinal (GI) surgeons, within liver surgery, the readers, to identify pre-defined anatomical landmarks in liver images processed by HS2, and assessment of landmark distance between CT and Holographic visualization (HV).

DETAILED DESCRIPTION:
This is a retrospective investigation of Computer Topographies (CTs)/ Holographic visualization based on CTs retrieved from patients with metastases in the liver from colorectal cancer.

The study consists of:

* Preparations at Day 0. The reader is not involved in the preparation
* Using of HS2 and evaluation at Day 1-2
* Calculation at Day 3.

The study will enroll eligible subject's images.

ELIGIBILITY:
Inclusion Criteria:

1. Livers with colorectal cancer liver metastasis
2. CTs from individuals 22 years or older
3. CTs retrieved from US hospitals
4. CTs from patients treated in the US
5. At least 1 visible liver lesion to complete detection of L1

Exclusion Criteria:

No exclusion criteria

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: US patients whose liver CT images will be used to create HVs.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2023-03-04 (Actual); Study Completion 2023-03-04 (Actual)

PRIMARY OUTCOMES:
Identification of all pre-defined landmarks. | 3 days
  All readers able to identify all pre-defined landmarks.

SECONDARY OUTCOMES:
Comparison between CT and HV distance. | 3 days
  Comparison between CT and HV distance in mm between a marker in a defined center of each portal landmark (difference less than 8.0 mm).
Comparison of image quality between CT and HV. | 3 days
  Comparison of image quality between CT and HV on a 5-graded scale (1=HV significantly poorer quality than CT, 2=HV somewhat poorer quality than CT, 3=HV as good as CT, 4=HV somewhat better than CT, 5=HV significantly better than CT). More than 50% should be scored as HV as good as CT or better. All five readers scoring 3 or higher.
Evaluate ease of use. | 3 days
  Evaluate ease of use on a 5-graded scale (1=very difficult, 2=difficult, 3=neither difficult nor easy, 4=easy, 5=very easy). All five readers scoring 4 or 5.

CONTACTS AND LOCATIONS:
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States